CLINICAL TRIAL: NCT06415357
Title: Adapting mHealth Interventions to Improve Self-management of HIV and Substance Use Among Emerging Adults in Zambia
Brief Title: Zambia Healthy Choices Project for Emerging Adults Living With HIV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Zambia (Other)
Responsible Party: Principal Investigator, Bo Wang, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001496; 1R34DA059935 (NIH)
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Pre-Exposure Prophylaxis
Keywords: Pre-Exposure Prophylaxis (PrEP); HIV Prevention; mHealth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard ART counseling, mHC, and MTM (Experimental): Participants in this arm will receive standard ART counseling, followed by two mHealth interventions (mHC and MTM) to improve PrEP uptake and adherence.
  Interventions: Behavioral: Mobile Healthy Choices (mHC); Behavioral: Motivational Text Messaging (MTM); Behavioral: Standard ART Counseling
- Standard ART counseling and mHC (Experimental): Participants in this arm will receive standard ART counseling, followed by one mHealth intervention (mHC) to improve PrEP uptake and adherence.
  Interventions: Behavioral: Mobile Healthy Choices (mHC); Behavioral: Standard ART Counseling
- Standard ART counseling and MTM (Experimental): Participants in this arm will receive standard ART counseling, followed by one mHealth intervention (MTM) to improve PrEP uptake and adherence.
  Interventions: Behavioral: Motivational Text Messaging (MTM); Behavioral: Standard ART Counseling
- Standard ART counseling (Active Comparator): Participants in this arm will receive standard ART counseling.
  Interventions: Behavioral: Standard ART Counseling

INTERVENTIONS:
Behavioral: Mobile Healthy Choices (mHC) — mHC is a four-session computer-delivered intervention based on the Information-Motivation-Behavioral (IMB) model and socioecological model (SEM). Using motivational interviewing, it tailors content to participants' responses. Sessions 1 and 2 focus on HIV self-management and alcohol reduction, gauging importance, confidence, and goals. Strengths, barriers, resources, and strategies are explored. Sessions 3 and 4 review goals, reinforce importance, confidence, and motivation, and strategize behavior maintenance. Over two months, participants engage in goal-oriented sessions, promoting sustained behavior change.
  Arms: Standard ART counseling and mHC; Standard ART counseling, mHC, and MTM
Behavioral: Motivational Text Messaging (MTM) — Text messages with motivational statements will be sent to participants based on their readiness to change, as assessed during mHC session 1. The statements promoting HIV self-management and alcohol use reduction will be derived from an MTM library written by Zambian young people living with HIV. MTM will be delivered to participants daily for two months and weekly for an additional four months at a time that a participant prefers.
  Arms: Standard ART counseling and MTM; Standard ART counseling, mHC, and MTM
Behavioral: Standard ART Counseling — All participants will receive one-on-one, face-to-face in clinic. Standard ART counseling includes the management and treatment of HIV, reproductive health, substance abuse, and mental health. They will also be counseled about treatment adherence and side-effect management.

SUMMARY:
This project will develop and implement a multi-component intervention using mobile health technology to improve HIV self-management and reduce substance use. Specifically, the investigators will adapt Healthy Choices (HC) to develop mobile HC (mHC) and develop Motivational text messaging (MTM) for Zambian emerging adults living with HIV.

ELIGIBILITY:
Zambian emerging adults living with HIV

Inclusion Criteria:

* Aged between 18 and 24 years
* Report visual analogue scale showing <80% medication adherence in the last month AND problematic/risky alcohol use in the last month
* Speak English, Nyanja, or Bemba

Exclusion Criteria:

* Have a serious cognitive or psychiatric problem that would compromise ability to provide informed consent
* currently enrolled in another HIV intervention study

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Intervention Acceptability: System Usability Score (SUS) | Month 3
  SUS is a 10-item, 5-point Likert scale for subjective assessment of usability. Each item ranges from 1 to 5. Depending on the item, the score is calculated by subtracting either one from the user response or the user response from 5. Then, the score for each item will be summed and multiplied by 2.5 for the total score. The overall SUS scores range from 0 to 100. A score of > 50 indicates that the technology-based interventions are acceptable.
Intervention Acceptability: System Usability Score (SUS) | Month 6
  SUS is a 10-item, 5-point Likert scale for subjective assessment of usability. Each item ranges from 1 to 5. Depending on the item, the score is calculated by subtracting either one from the user response or the user response from 5. Then, the score for each item will be summed and multiplied by 2.5 for the total score. The overall SUS scores range from 0 to 100. A score of > 50 indicates that the technology-based interventions are acceptable.
Intervention Acceptability: Client Satisfaction Questionnaire (CSQ-8) | Month 3
  CSQ-8 is an 8-item, 4-point Likert scale measuring the construct of global intervention satisfaction. The total possible composite score ranges from 8 to 32, with higher scores indicating greater acceptability.
Intervention Acceptability: Client Satisfaction Questionnaire (CSQ-8) | Month 6
  CSQ-8 is an 8-item, 4-point Likert scale measuring the construct of global intervention satisfaction. The total possible composite score ranges from 8 to 32, with higher scores indicating greater acceptability.
Intervention Acceptability: Exit Interview | Month 3
  Participants will be invited to share their experiences with mHC and MTM, including feedback on acceptability, ease of use, suggestions for improvement, and impact on ART adherence and alcohol use reduction.
Intervention Feasibility: Participant Retention | Baseline to Month 6
  Intervention feasibility will be assessed based on participant retention at Month 6. The retention rate can range from 70 to 90%, with a retention rate of over 85% deemed the minimum criterion for feasibility.
Intervention Feasibility: Number of Responses to MTM | Baseline to Month 6
  Intervention feasibility will be evaluated by the total number of responses to MTM.
Intervention Feasibility: Number of mHC Sessions Completed | Baseline to Month 6
  Intervention feasibility will be evaluated by the number of completed intervention sessions.
ART Adherence: Visual Analog Scale | Baseline, Month 3, and Month 6
  ART adherence will be assessed through the Young Adult Adherence Interview via computer-assisted self-interview (CASI) survey, which contains a visual analog scale (VAS) ranging from 0 to 100. Higher percentages on the VAS indicate greater adherence to ART.
ART Adherence: Self-Reported Adherence | Baseline, Month 3, and Month 6
  ART adherence will be evaluated through self-reported adherence over the past four weeks via a CASI survey. Participants will rate their adherence on a scale ranging from 0 to 100%, with higher percentages indicating better adherence to ART.
ART Adherence: Dried Blood Spot (DBS) Testing | Baseline, Month 3, and Month 6
  ART adherence will be evaluated by examining the HIV viral load in DBS. Maintaining a viral load of less than 200 copies/ml will indicate adherence to ART.
Alcohol Use: The Timeline Followback (TLFB) Interview | Baseline, Month 3, and Month 6
  Alcohol use will be assessed using the TLFB interview. Using a calendar, participants will be asked to provide estimates of their daily drinking over the last 30 days, as well as the max number of drinks in a one-week period, the number of heavy drinking days, the number of standard drinks in 30 days, and binge drinking.

SECONDARY OUTCOMES:
Information: HIV Knowledge | Baseline, Month 3, and Month 6
  HIV transmission risk awareness will be evaluated through an 18-item HIV Knowledge Questionnaire. Total possible composite scores range from 0 to 18, with higher scores indicating a higher level of HIV knowledge.
Information: ART Knowledge | Baseline, Month 3, and Month 6
  ART knowledge will be evaluated through a 21-item HIV Treatment Knowledge Questionnaire. Total possible composite scores range from 0 to 21, with higher scores indicating a higher level of ART knowledge.
Motivation: Rollnick's Readiness Ruler | Baseline, Month 3, and Month 6
  Intentions to improve HIV self-management and alcohol consumption behaviors will be evaluated using the 5-item Rollnick's Readiness Ruler. Each item ranges from 0 to 10, with higher scores indicating a greater readiness for change.
Motivation: Decisional Balance for Problem Behavior | Baseline, Month 3, and Month 6
  Attitudes toward risk behaviors will be assessed using the 32-item Decisional Balance for Problem Behavior scale. This 5-point Likert scale evaluates the perceived pros and cons of engaging in risk behaviors
Behavioral Skills: Self-Efficacy | Baseline, Month 3, and Month 6
  Behavioral skills in HIV self-management will be assessed using a 5-item adapted version of the Self-Efficacy for Health Promotion and Risk Reduction Questionnaire. This 5-point Likert scale measures confidence levels (score range: 5-25), with higher scores indicating greater confidence in HIV self-management tasks.
STI Diagnosis: Number of participants who are diagnosed with syphilis, gonorrhea, or chlamydia | Baseline and Month 6
  Syphilis testing will employ a treponemal test with rapid plasma reagin (RPR), while gonorrhea and chlamydia testing will utilize pooled urine, oropharyngeal, and rectal swabs.
Sexual Risk | Baseline, Month 3, and Month 6
  Sexual risk will be assessed using TLFB interview via CASI, capturing sexual behavior over the past 30 days, such as condom usage and the number of sexual partners.
Drug Use: Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) | Baseline, Month 3, and Month 6
  Drug use will be assessed with ASSIST, which is a questionnaire to identify substance use health risks and disorders, with each item scored from 0 to 12. The total score ranges up to 24, with higher scores indicating greater risk based on current substance use patterns.
Drug Use: Alcohol Use Disorder Identification Text (AUDIT-C) | Baseline, Month 3, and Month 6
  Alcohol use will be assessed by using AUDIT-C to identify individuals with hazardous drinking habits or alcohol use disorders. Each item scores from 0 to 4, with 0 indicating no alcohol consumption. The total score maxes out at 12, with higher scores suggesting greater risks of harm.
Mental health: Brief Symptom Inventory (BSI-18) | Baseline, Month 3, and Month 6
  Mental health will be evaluated with BSI-18. This 18-item questionnaire utilizes a 5-point Likert scale to gauge psychological distress. Scores range up to 72, with higher scores indicating a higher level of psychological distress.
Social support: Social Provision Scale | Baseline, Month 3, and Month 6
  Social support will be evaluated using the Social Provision Scale. This 5-point Likert scale, 13-item survey assesses the availability of social support, such as emotional, information, and instrumental support, as well as companionship and social isolation. Scores range up to 65, with higher scores indicating more extensive availability of social support.
HIV stigma: Shortened Version of Berger's Stigma Scale | Baseline, Month 3, and Month 6
  HIV-related stigma will be evaluated using the 10-item Berger's Stigma Scale. This scale, based on a 4-point Likert scale, assesses the stigma perceived by people living with HIV. The score can range from 10 to 40, with a higher score indicating greater perceived stigma associated with HIV.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Wang, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wises to access the data.

REFERENCES:
- [Background] Chenneville T, Machacek M, St John Walsh A, Emmanuel P, Rodriguez C. Medication Adherence in 13- to 24-Year-Old Youth Living With HIV. J Assoc Nurses AIDS Care. 2017 May-Jun;28(3):383-394. doi: 10.1016/j.jana.2016.11.002. Epub 2016 Nov 11. PMID 27931753
- [Background] Nabukeera-Barungi N, Elyanu P, Asire B, Katureebe C, Lukabwe I, Namusoke E, Musinguzi J, Atuyambe L, Tumwesigye N. Adherence to antiretroviral therapy and retention in care for adolescents living with HIV from 10 districts in Uganda. BMC Infect Dis. 2015 Nov 14;15:520. doi: 10.1186/s12879-015-1265-5. PMID 26573923
- [Background] St Clair-Sullivan N, Mwamba C, Whetham J, Bolton Moore C, Darking M, Vera J. Barriers to HIV care and adherence for young people living with HIV in Zambia and mHealth. Mhealth. 2019 Sep 30;5:45. doi: 10.21037/mhealth.2019.09.02. eCollection 2019. PMID 31620472
- [Background] Williams EC, Hahn JA, Saitz R, Bryant K, Lira MC, Samet JH. Alcohol Use and Human Immunodeficiency Virus (HIV) Infection: Current Knowledge, Implications, and Future Directions. Alcohol Clin Exp Res. 2016 Oct;40(10):2056-2072. doi: 10.1111/acer.13204. Epub 2016 Sep 22. PMID 27696523
- [Background] Denison JA, Packer C, Stalter RM, Banda H, Mercer S, Nyambe N, Katayamoyo P, Mwansa JK, McCarraher DR. Factors Related to Incomplete Adherence to Antiretroviral Therapy among Adolescents Attending Three HIV Clinics in the Copperbelt, Zambia. AIDS Behav. 2018 Mar;22(3):996-1005. doi: 10.1007/s10461-017-1944-x. PMID 29103190
- [Background] Tarantino N, Lowery A, Brown LK. Adherence to HIV Care and Associated Health Functioning among Youth Living with HIV in Sub-Saharan Africa. AIDS Rev. 2020 Jul 8;22(2):93-102. doi: 10.24875/AIDSRev.20000101. PMID 32180589
- [Background] Scott-Sheldon LA, Carey KB, Cunningham K, Johnson BT, Carey MP; MASH Research Team. Alcohol Use Predicts Sexual Decision-Making: A Systematic Review and Meta-Analysis of the Experimental Literature. AIDS Behav. 2016 Jan;20 Suppl 1(0 1):S19-39. doi: 10.1007/s10461-015-1108-9. PMID 26080689
- [Background] Hendershot CS, Stoner SA, Pantalone DW, Simoni JM. Alcohol use and antiretroviral adherence: review and meta-analysis. J Acquir Immune Defic Syndr. 2009 Oct 1;52(2):180-202. doi: 10.1097/QAI.0b013e3181b18b6e. PMID 19668086
- [Background] Mulawa MI, LeGrand S, Hightow-Weidman LB. eHealth to Enhance Treatment Adherence Among Youth Living with HIV. Curr HIV/AIDS Rep. 2018 Aug;15(4):336-349. doi: 10.1007/s11904-018-0407-y. PMID 29959649
- [Background] Doyle AM, Bandason T, Dauya E, McHugh G, Grundy C, Dringus S, Dziva Chikwari C, Ferrand RA. Mobile Phone Access and Implications for Digital Health Interventions Among Adolescents and Young Adults in Zimbabwe: Cross-Sectional Survey. JMIR Mhealth Uhealth. 2021 Jan 13;9(1):e21244. doi: 10.2196/21244. PMID 33439136
- [Background] Ramsey SE, Ames EG, Uber J, Habib S, Clark S, Waldrop D. A Preliminary Test of an mHealth Facilitated Health Coaching Intervention to Improve Medication Adherence among Persons Living with HIV. AIDS Behav. 2021 Nov;25(11):3782-3797. doi: 10.1007/s10461-021-03342-5. Epub 2021 Jun 12. PMID 34117965
- [Background] Cooper V, Clatworthy J, Whetham J, Consortium E. mHealth Interventions To Support Self-Management In HIV: A Systematic Review. Open AIDS J. 2017 Nov 21;11:119-132. doi: 10.2174/1874613601711010119. eCollection 2017. PMID 29290888
- [Background] Hutton A, Prichard I, Whitehead D, Thomas S, Rubin M, Sloand E, Powell TW, Frisch K, Newman P, Goodwin Veenema T. mHealth Interventions to Reduce Alcohol Use in Young People: A Systematic Review of the Literature. Compr Child Adolesc Nurs. 2020 Sep;43(3):171-202. doi: 10.1080/24694193.2019.1616008. Epub 2019 Jun 13. PMID 31192698
- [Background] Garofalo R, Kuhns LM, Hotton A, Johnson A, Muldoon A, Rice D. A Randomized Controlled Trial of Personalized Text Message Reminders to Promote Medication Adherence Among HIV-Positive Adolescents and Young Adults. AIDS Behav. 2016 May;20(5):1049-59. doi: 10.1007/s10461-015-1192-x. PMID 26362167
- [Background] Suffoletto B, Chung T, Muench F, Monti P, Clark DB. A Text Message Intervention with Adaptive Goal Support to Reduce Alcohol Consumption Among Non-Treatment-Seeking Young Adults: Non-Randomized Clinical Trial with Voluntary Length of Enrollment. JMIR Mhealth Uhealth. 2018 Feb 16;6(2):e35. doi: 10.2196/mhealth.8530. PMID 29453191
- [Background] Horvath KJ, Smolenski D, Amico KR. An empirical test of the information-motivation-behavioral skills model of ART adherence in a sample of HIV-positive persons primarily in out-of-HIV-care settings. AIDS Care. 2014 Feb;26(2):142-51. doi: 10.1080/09540121.2013.802283. Epub 2013 Jun 3. PMID 23724908
- [Background] Amico KR, Barta W, Konkle-Parker DJ, Fisher JD, Cornman DH, Shuper PA, Fisher WA. The information-motivation-behavioral skills model of ART adherence in a Deep South HIV+ clinic sample. AIDS Behav. 2009 Feb;13(1):66-75. doi: 10.1007/s10461-007-9311-y. Epub 2007 Sep 18. PMID 17876697
- [Background] Naar-King S, Outlaw AY, Sarr M, Parsons JT, Belzer M, Macdonell K, Tanney M, Ondersma SJ; Adolescent Medicine Network for HIV/AIDS Interventions. Motivational Enhancement System for Adherence (MESA): pilot randomized trial of a brief computer-delivered prevention intervention for youth initiating antiretroviral treatment. J Pediatr Psychol. 2013 Jul;38(6):638-48. doi: 10.1093/jpepsy/jss132. Epub 2013 Jan 28. PMID 23359664
- [Background] Murphy DA, Chen X, Naar-King S, Parsons JT; Adolescent Trials Network. Alcohol and marijuana use outcomes in the Healthy Choices motivational interviewing intervention for HIV-positive youth. AIDS Patient Care STDS. 2012 Feb;26(2):95-100. doi: 10.1089/apc.2011.0157. Epub 2011 Dec 22. PMID 22191456